CLINICAL TRIAL: NCT01780805
Title: Second Young Adult Naturalistic Alcohol Study (YANAS-2)
Brief Title: Second Young Adult Naturalistic Alcohol Study
Acronym: YANAS-2
Status: Completed | Type: Observational
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 1209010754; R03AA022232 (NIH)
Record Dates: First submitted 2013-01-24; First posted 2013-01-31 (Estimated); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Young Adult Alcohol Drinking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Young adult alcohol drinkers: Young adults between the ages of 21-25 who regularly drink alcohol

SUMMARY:
This study involves completion of questionnaires, computer-based cognitive tasks and an alcohol drinking session. Participation in this study consists of an initial, in-person screening appointment, 4 brief daily appointments at the research office, an alcohol drinking session at a local bar and a follow-up appointment 1-3 days after the alcohol drinking session.

Participants who are found to be eligible in the screening phase will then complete a daily appointment for 4 days out of a 5-day period (i.e., there will be 1 day out of the 5 on which they will not attend an appointment). Each appointment will last 20 minutes, on average and consist of a questionnaire and computer-based cognitive task. On the day of the fourth appointment, participants will complete an alcohol drinking session. The alcohol drinking session begins at 4pm and lasts until at least midnight.

Participants in this study will be young adults between the ages of 21-25, who regularly drink alcohol and are not currently seeking treatment for alcohol use. Seventy-two participants will complete this study.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 21-25.
* Be able to read English and complete study evaluations.
* Drink alcohol on a regular basis

Exclusion Criteria:

No participant may:

* Be seeking treatment for alcohol or other addictive behaviors or have been in inpatient or intensive outpatient treatment within the past 12 months.
* Provide two positive breath alcohol concentration (BAC) readings (i.e., > 0.00%) at any of the following times: in-person screening, a pre-session screening, or at the outset of an alcohol self-administration session. After participants blow their first positive BAC, they will be allowed to reschedule and participate at another time, however if they blow a second positive BAC, they will be excluded from this study and offered referrals for alcohol treatment.
* Have positive urine screen results at the in-person screening or pre-session screening on the day of an alcohol self-administration session for opiates, cocaine, phencyclidine, amphetamines, methamphetamine, barbiturates, methadone or benzodiazepines.
* A woman who is pregnant, nursing, or refuses to use a reliable method of birth control.
* Fail to perform at a normative level at screening on any of the four cognitive and psychomotor tasks administered in this study. Participants must perform within two standard deviations of the mean from the samples in relevant prior studies
* Perform computer tasks initially administered at baseline in either a random or inordinately slow fashion
* A body mass index lower than 18.5 or greater than 35.

Ages: 21 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy young adults between the ages of 21-25 years of ago who regularly drink alcohol and are not currently seeking treatment for alcohol.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2013-01; Primary Completion 2015-11 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Peak estimated blood alcohol concentration | During a 3-hour alcohol drinking period

SECONDARY OUTCOMES:
Number of alcoholic drinks consumed | During a 3-hour alcohol drinking period

OTHER OUTCOMES:
Self-reported drinks per drinking day | 6- and 12-month follow-ups after alcohol drinking session
Self-reported frequency of heavy drinking days | 6- and 12-month follow-up after alcohol drinking session

CONTACTS AND LOCATIONS:
Overall Officials: Robert F Leeman, Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States